CLINICAL TRIAL: NCT00488592
Title: Efficacy of Peptide (WT1) and Peptide(PRI) Vaccination for Patients With Low Risk Myeloid Malignancies
Brief Title: Peptide Vaccinations to Treat Patients With Low-Risk Myeloid Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070159; 07-H-0159 (Other: National Heart Lung and Blood Institute); NCT00499772 (obsolete NCT alias)
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2014-06

CONDITIONS: Myelodysplastic Syndrome (MDS); Acute Myeloid Leukemia (AML); Chronic Myeloid Leukemia (CML)
Keywords: Myelodysplastic Syndrome (MDS); Acute Myeloid Leukemia (AML); Chronic Myeloid Leukemia (CML); Wilm's Tumor-1; Proteinase-3; Myelodysplastic Syndrome; MDS; Acute Myeloid Leukemia; AML; Chronic Myeloid Leukemia; CML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — WT1 (126-134), human; Peptides; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Colony-Stimulating Factors; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers (Experimental): Subjects were given 6 subcutaneous injects of PR1:169-177 in "Montanide" adjuvant and 6 subcutaneous injections of WT1:126-134 in "Montanide" adjuvant at 2 weekly intervals. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
  Interventions: Biological: WT1:126-134; Biological: PR1:169-177 Peptide; Drug: GM-CSF (Sargramostim); Biological: Montanide adjuvant

INTERVENTIONS:
Biological: WT1:126-134 — Subjects were given 6 doses of PR1:169-177 in "Montanide" adjuvant and 6 doses of WT1:126-134 in "Montanide" adjuvant at 2 weekly intervals. The peptides were injected in the deep subcutaneous tissue of the anterior abdominal wall, the thighs or the upper arms near the deltoid region. The sites of injection were rotated every 2 weeks. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
  Other Names: Wilms' tumor 1: 126-134 (WT1:126-134) Peptide
Biological: PR1:169-177 Peptide — Subjects were given 6 doses of PR1:169-177 in montanide adjuvant and 6 doses of WT-1:126-134 in Montanide adjuvant at 2 weekly intervals. The peptides were injected in the deep subcutaneous tissue of the anterior abdominal wall, the thighs or the upper arms near the deltoid region. The sites of injection were rotated every 2 weeks. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
  Other Names: peptide (PR1:169-177)
Drug: GM-CSF (Sargramostim) — Subjects were given 6 doses of PR1:169-177 in montanide adjuvant and 6 doses of WT-1:126-134 in Montanide adjuvant at 2 weekly intervals. The peptides were injected in the deep subcutaneous tissue of the anterior abdominal wall, the thighs or the upper arms near the deltoid region. The sites of injection were rotated every 2 weeks. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
  Other Names: granulocyte macrophage colony- stimulating factor (GM-CSF)
Biological: Montanide adjuvant — Subjects were given 6 doses of PR1:169-177 in montanide adjuvant and 6 doses of WT-1:126-134 in Montanide adjuvant at 2 weekly intervals. The peptides were injected in the deep subcutaneous tissue of the anterior abdominal wall, the thighs or the upper arms near the deltoid region. The sites of injection were rotated every 2 weeks. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.

SUMMARY:
This study will test the safety and effectiveness of two vaccines on slowing disease progression, improving blood counts, reducing the need for transfusions of blood and platelets, or achieving remission in patients with myelodysplastic syndrome (MDS, also known as myelodysplasia), acute myeloid leukemia (AML) or chronic myeloid leukemia (CML). The vaccines consist of peptides (parts of proteins) found in MDS, AML and CML stem cells, combined with a substance called "MontanideTM". They are administered with granulocyte- macrophage colony- stimulating factor (GM-CSF). The Montanide and the GM-CSF help the immune system respond to the vaccines.

People 18 years of age or older with MDS, AML or CML may be eligible for this study.

Participants receive six injections of the vaccines, one dose every other week for a total of 10 weeks. The injections are given in the upper arm, upper leg, or abdomen. A separate injection of GM-CSF is given in the same area as the vaccine injections. Subjects are observed for 2 hours after the first vaccination and at least 30 minutes after each subsequent vaccination for allergic reactions. In addition to the vaccination, subjects undergo the following:

* History and physical exam, chest x-ray, blood tests and bone marrow aspirate and biopsy before starting the vaccinations.
* Safety monitoring during vaccine administration (every other week for 10 weeks) with blood tests and check of vital signs.
* Follow-up safety monitoring (weeks 12 and 16) with blood tests every visit, chest x-ray at week 12 and bone marrow biopsy visit 16.

DETAILED DESCRIPTION:
Leukemias and the related disorders myelodysplastic syndrome and myeloproliferative diseases represent a wide group of bone marrow stem cell malignancies. Some patients can be cured with chemotherapy or by allogeneic stem cell transplantation. However standard treatment approaches are not effective for patients who become refractory to chemotherapy, those who relapse after transplantation and those with progressive disease. The management of such patients remains unsatisfactory and requires new treatment approaches other than chemotherapy.

The immunological graft-versus-leukemia (GVL) effect seen after allogeneic stem cell transplantation suggests that stimulating the patient's own T cell responses to MDS and leukemia with a vaccine might also retard disease progression and even achieve disease remissions. Peptide (WT1) and peptide (PR1) were identified as target antigens because both antigens are highly expressed by cluster of differentiation 34 (CD34) plus stem cells of most patients with myeloid malignancies but not by normal marrow cells. An immunotherapeutic approach to vaccinate against PR1 and WT1 antigens could induce T cell response against MDS and leukemic cells while sparing normal cells and by using a combination of two antigens the risk of disease escape by antigen down regulation should be further diminished. Indeed in a safety study of one dose of a combination of peptide (PRl) and (WT1) vaccination, we demonstrated that immunological response against one or both vaccines could be induced in all subjects who were vaccinated. This immunological response was associated with a transient reduction in the leukemia burden. Furthermore the vaccine combination was well tolerated.

Therefore we propose this Phase II trial, the third in a series of planned peptide vaccine research protocols, which will evaluate the safety and efficacy associated with an immunotherapy approach using two peptide vaccines, namely PR 1 : 169- 177 and WT-1: 126-1 34 in Montanide adjuvant, administered concomitantly with GM-CSF (Sargramostim), every 2 weeks for 10 weeks (6 doses WT1 plus 6 doses PRl plus GM-CSF) in select patients diagnosed with MDS, AML or CML. Subjects with immunological response to one or both peptide vaccines will have the option of receiving an additional 6 boosters of the WT-1:126-135 and PR1:169-177 peptide vaccines at 3 monthly intervals.

The primary objective will be to evaluate the efficacy and toxicity associated with 6 doses of a combination of WT-1: 126-134 and PRl: 169-177 peptide vaccines in Montanide adjuvant administered concomitantly with GMCSF (Sargramostim) in selected patients with myeloid malignancies (MDS, AML, CML).

The primary endpoint will be immune response (studying changes in the frequencies of circulating PR1 and WT1 specific T cells) which will serves as a surrogate for evaluating for the efficacy of the study.

Secondary Endpoints will include changes in marrow blast cells, blood counts, transfusion dependence, time to disease progression and survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosed with MDS (B subtypes Refractory anemia (RA), Refractory anemia with ring sideroblasts (RARS) -Low Risk) (MDS with 5q- must have failed lenalidomide or been ineligible to receive it)

OR

Diagnosed with AML and in complete remission within 5 years of treatment with less than 5% marrow blasts

OR

Diagnosed with CML in chronic phase

Unsuitable for stem cell transplantation (SCT) (age over sixty or unavailability of a fully-matched donor)

or

made an informed decision not to undergo the transplant procedure

or

are between 6 months 3 years following allogeneic SCT and fulfill the following criteria:

100% donor engraftment,

Less than 5% blasts in marrow

normal marrow cellularity

Human leukocyte antigen (HLA-A020 1) positive at one allele

Ages 18-85 years old

Off all lympho-ablative chemotherapeutic agents

EXCLUSION CRITERIA:

* Hypoplastic MDS
* Relapsed AML
* CML in accelerated phase or blast crisis
* Hypocellular bone marrow (less than 20%)
* History of Wegener's granulomatosis
* Serologic antibody against proteinase-3 (ANCA positive)
* Previous allergic reaction to Montanide Adjuvant
* Positive test for HIV
* Treatment with systemic corticosteroids or immunosuppressants within 14 days prior to study entry
* Co-morbidity of such severity that it would preclude the patient's ability to tolerate protocol therapy
* Predicted survival less than 28 days
* Pregnant or breast feeding (All female patients must have a urine pregnancy test within 1 week prior to vaccine administration)
* Unwilling to practice abstinence or effective contraception (men and women) during the study period.
* Enrolled in another drug or vaccine clinical trial during the study period
* Inability to comprehend the investigational nature of the study and provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minocher Battiwalla, MD, Principal Investigator — National Institutes of Health- NHLBI
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rezvani K, Yong AS, Mielke S, Jafarpour B, Savani BN, Le RQ, Eniafe R, Musse L, Boss C, Kurlander R, Barrett AJ. Repeated PR1 and WT1 peptide vaccination in Montanide-adjuvant fails to induce sustained high-avidity, epitope-specific CD8+ T cells in myeloid malignancies. Haematologica. 2011 Mar;96(3):432-40. doi: 10.3324/haematol.2010.031674. Epub 2010 Dec 6. PMID 21134985
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2007-H-0159.html

RESULTS

PARTICIPANT FLOW:
Groups:
- PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers: Participants were given subcutaneous 6 injections of PR1:169-177 in "Montanide" adjuvant and 6 doses of WT1:126-134 in "Montanide" adjuvant at 2 weekly intervals. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
Period: Overall Study
Arm/Group | PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers
Started | 10 (10 subjects were accrued)
Completed | 7 (7 completed the initial series of 6 vaccinations)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 1
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Inducing or Boosting of a Cellular Immune Response
Description: Number of participants diagnosed with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML) or chronic myeloid leukemia (CML) who experienced an inducing or boosting of a cellular immune response following Wilm's Tumor 1 (WT1) and PR1 vaccine.
  A T-cell immune response was considered positive if the frequencies of interferon (IFN-γ+) cluster of differentiation (CD8+) T cells in peptide-stimulated peripheral bloody mono-nucleated cells (PBMCs) were 2-fold or more higher than the frequencies of interferon (IFN-γ+) CD8+ T cells in unstimulated PBMCs and if there was a minimum of 0.05% Interferon (IFNγ+) CD8+ T cells (after subtracting the frequencies of interferon (IFNγ+) CD8+ T cells in unstimulated PBMCs). A significant vaccine-induced CD8+ T-cell response was defined as the emergence of detectable PR1 or WT1-specific CD8+ T cells when the pre-study analysis found no response, or a 2-fold increase in frequencies when responses were present before vaccination.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers
Number analyzed (Participants) | 7
participants
  Cellular immune response | 5
  No cellular immune response | 2

2. Secondary Outcome: Number of Participants Who Experienced a Hematological Response
Description: Number of participants diagnosed with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML) or chronic myeloid leukemia (CML) who experienced a hematological response following Wilm's Tumor (WT1) and PR1 peptide vaccine.
  Hematological response is defined by reduction in marrow blast cells, changes in blood counts.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | PR1/WT1 Vaccine Response in Participants With Low-Risk Myeloid Cancers
Number analyzed (Participants) | 7
participants | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- PR1/WT1 Vaccine Response in Participants With Leukemias: Participants were given subcutaneous 6 injections of PR1:169-177 in "Montanide" adjuvant and 6 doses of WT1:126-134 in "Montanide" adjuvant at 2 weekly intervals. GM-CSF (Sargramostim) was co administered with each vaccine dose. Subjects with immunological response to one or both peptide vaccines had the option of receiving a maximum of 6 additional boosters of the WT-1:126-134 and PR1:169-177 peptide vaccines at 3 monthly intervals.
Arm/Group | PR1/WT1 Vaccine Response in Participants With Leukemias
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR1/WT1 Vaccine Response in Participants With Leukemias (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — found to be related to relapsed disease
Upper Respiratory Infection (Infections and infestations) | 1 (1) — Bronchoscopy positive for staph and strep
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR1/WT1 Vaccine Response in Participants With Leukemias (N=10)
decreased hemoglobin (Blood and lymphatic system disorders) | 1 (1)
back pressure (Immune system disorders) | 2 (2)
fatigue (General disorders) | 1 (1)
lightheadness (General disorders) | 1 (1)
malaise (General disorders) | 1 (1)
rigors (General disorders) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 4 (4)
indigestion (Gastrointestinal disorders) | 1 (1)
loose stools (Gastrointestinal disorders) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes